CLINICAL TRIAL: NCT05919927
Title: Effects of Type II Diabetes on Cognitive Functions in Middle-aged Patients
Brief Title: Diabetes and Cognitive Functions in Middle Age
Acronym: DBC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: TAUCH
Record Dates: First submitted 2016-11-07; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Impairment; Hyperglycemia; Hypoglycemia; Mood
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type II diabetes patients: Neuropsychological examination is done and medical information is gathered from the medical records.
- Healthy controls: Neuropsychological examination, medical examination and laboratory tests.

SUMMARY:
This study will examine the effects of type II diabetes on cognitive functions and mood in middle-aged patients. In addition, the association between cognitive functions and glycemic controls is studied in patients. Sixty patients and sixty healthy controls will be recruited and assessed by a multiprofessional team (neuropsychologist, physician).

DETAILED DESCRIPTION:
Sixty patients with type 2 diabetes will be recruited from the Tampere Diabetes outpatient clinic. Inclusion criteria for the patients are type 2 diabetes diagnosis, diabetes medication and age 35-65. Exclusion criteria are type 1 diabetes, hypothyreosis, neurological or psychiatric disorder, substance abuse and serious diabetes complications. Sixty healthy control persons are recruited from the personnel and occupational health care. Exclusion criteria for controls are type 1 or 2 diabetes, hypothyreosis, neurological or psychiatric disease and substance abuse.

A comprehensive neuropsychological assessment is made to all participants.The assessment consists of standardized neuropsychological tests, questionnaires and interview. Domains assessed include attention, executive functions, memory, information processing speed, general cognitive functioning, depressive symptoms, anxiety and fatigue. Medical information (such as glycated hemoglobin and blood pressure) from the patients is gathered from the medical records. Corresponding information from the control participants is gathered with medical examinations including laboratory tests. Informed consent is taken from all participants.

This study will examine the difference in cognitive functions between healthy controls and middle-aged patients with type 2 diabetes. There is evidence from previous studies that type 2 diabetes is related to an increased risk of dementia, but the association between diabetes and cognition at younger ages is less studies. The difference in mood and fatigue is also studied between the groups. In addition, the association between glycated hemoglobin level and cognitive functions is examined in patients, as poor glycemic control has been implicated to impact on cognitive decline in previous studies. Finally, the association between history of hypoglycemic episodes and cognition is studied.

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes, age between 35-65 years

Exclusion Criteria:

* hypothyreosis, previous neurological diseases

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type II diabetes patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Adult Intelligence Scale-test | 1 day.
  Wechsler Adult Intelligence Scale-test and its z-score. Average performance differences in this cognitive test are compared between healthy controls and patients with type 2 diabetes using SPSS-program.
Continuous Performance test | 1 day.
  Continuous Performance test and its z-score. Average performance differences in this cognitive test are compared between healthy controls and patients with type 2 diabetes using SPSS-program.
Rey-Osterrieth Complex Figure test | 1 day.
  Rey-Osterrieth Complex Figure test and its z-score. Average performance differences in this cognitive test are compared between healthy controls and patients with type 2 diabetes using SPSS-program.
Sum score of the Z-scores of the performed standardized neuropsychological tests | 1 day.
  Sum score of the Z-scores of the performed standardized neuropsychological tests (Wechsler Adult Intelligence Scale, Continuous Performance test and Rey-Osterrieth Complex Figure test). Average performances evaluated by the differences in these sum scores are compared between healthy controls and patients with type 2 diabetes using SPSS-program.

CONTACTS AND LOCATIONS:
Overall Officials: Mervi Jehkonen, PhD, Principal Investigator — Tampere University
Locations (1):
- Tampere University Hospital, Tampere, Finland